CLINICAL TRIAL: NCT04107402
Title: Prospective Evaluation of PLatelets Acetyl-CoA Carboxylase Phosphorylation State in SEPtic Shock Patients. Impact of Platelets Metabolism to Inflammatory Response.
Brief Title: PLatelets Acetyl-CoA Carboxylase Phosphorylation State in SEPtic Shock
Acronym: PLACCSEPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PLACCSEPS; 2018/11DEC/469 (Other: CEHF)
Record Dates: First submitted 2019-04-11; First posted 2019-09-27 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Septic Shock; Platelet Signal Processing Defect; Inflammatory Response; Disseminated Intravascular Coagulation; Covid19; Neutrophil Extracellular Trap Formation
Keywords: Septic shock; Platelets; Acetyl CoA Carboxylase
MeSH Terms: conditions — Shock, Septic; Platelet Signal Processing Defect; Disseminated Intravascular Coagulation; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Septic shock (Experimental): Septic shock Patients admitted to the ICU
  Interventions: Other: Assessment of coagulopathy, Platelets activation and Platelets-Neutrophils interplay
- Control group (Other): Patients recruited at the central lab of the hospital, with matched age, gender and comorbidities
  Interventions: Other: Assessment of coagulopathy, Platelets activation and Platelets-Neutrophils interplay
- Covid-19 (Experimental): Covid-19 patients admitted to the ICU for Acute Respiratory Distress Syndrom with PaO2/FiO2 < 200
  Interventions: Other: Assessment of coagulopathy, Platelets activation and Platelets-Neutrophils interplay

INTERVENTIONS:
Other: Assessment of coagulopathy, Platelets activation and Platelets-Neutrophils interplay — Blood sample Urine Sample Pulmonary, hepatic and cardiac tissue from biopsy and autopsy
  Other Names: Inflammatory biomarkers; Coagulation assessment; Platelets activation state assessment; Neutrophils Extra-cellular trap assessment; Quantification and analysis of micro-thrombi; Platelets Acetyl-CoA Carboxylase phosphorylation analysis

SUMMARY:
Knowing the dramatic increase in thrombin generation during sepsis, our research hypothesis is that AMPK-induced ACC phosphorylation in platelets is increased and that this might modulate platelets metabolism and more particularly platelets inflammatory mediators content, coming from AA and lipids.

DETAILED DESCRIPTION:
Background

Sepsis, a systemic inflammatory reaction occurring in response to an infection, is a major public health problem and is recognized as the leading cause of death in the intensive care unit (ICU). This severe inflammatory reaction causes endothelial activation and dysfunction. This phenomenon is closely associated with the activation of coagulation cascade via exposure of tissue factor (TF) at endothelial cell surface. TF serves as an anchor for factors of coagulation VII and X allowing their activation. This results in thrombin (IIa) generation and fibrin production.

Thrombin is also a potent platelet agonist (activator) resulting in platelet activation and consumption. The pro-coagulant activity of activated platelets during sepsis enhances the formation of micro-thrombosis that impair organ perfusion and may lead to death. Thrombocytopenia is common and is a strong negative prognostic marker in septic shock patients.

Beyond coagulation, platelets are known to play a key role in inflammation and immune response. Platelets activation can be initiated by inflamed endothelium or circulatory inflammatory cytokines, which in turn, modulates the inflammatory and thrombotic response. Activated platelets interact with immune cells, like neutrophils. Furthermore, platelets can act as microbial "sensors" by expressing members of Toll-Like Receptors (TLRs) family, binding ligands from several infectious agents. Recent data highlight the interplay between platelets and neutrophils extracellular traps (NETs). Platelets facilitate NETs formation and, inversely, NETS activate platelets. NETs connect platelets, thrombosis, immune response and inflammation and therefore are of particular interest in the septic context.

Platelets express Acetyl-CoA carboxylase 1 (ACC1), which is the first step enzyme of lipogenesis. ACC Phosphorylation on Serine 79 by AMP-activated protein kinase (AMPK) leads to its inhibition and AMPK is activated by thrombin. We demonstrated that AMPK-ACC axis controls platelets phospholipids content, which influence TXA2 and dense granule release and, in turn, thrombus formation. TXA2 is generated from phospholipids containing arachidonic acid (AA). Alternatively, AA can be metabolized by lipooxygenase (LOX) pathway producing lipoxins (LX) and resolvin, which are rather involved in the resolution of inflammation. The relation between AMPK-ACC signalling and lipooxygenase pathway has never been investigated.

Research hypothesis

Knowing the dramatic increase in thrombin generation during sepsis, our research hypothesis is that AMPK-induced ACC phosphorylation in platelets is increased and that this might modulate platelets metabolism and more particularly platelets inflammatory mediators content, coming from AA and lipids.

Patients selection

Consecutive patients with septic shock admitted at Cliniques universitaires Saint-Luc, Brussels, will be included (experimental group)

Control group will correspond to healthy volunteers with matched age and gender, based on retrospective analysis of patients admitted in ICU for sepsis.

Exploratory control group will correspond to patients admitted in the intensive care unit without evidence of severe infection and severe systemic inflammatory response. Patients with neurological disorder and intoxication will be the target population.

Similar exclusion criteria will be the same in control groups than in the experimental group.

Material and methods

Type of study Prospective, monocentric, interventional study.

Blood sampling Blood samples will be collected after venous catheter insertion, within 48 hours after septic shock diagnosis.

The following samples will be taken during the procedure:

* Coagulation including (INR, TCA, TT, PTT, Fibrinogen, DDimers) (1 green TUBE of 3 ml)
* Multiplate analysis (1 orange TUBE of 3 ml)
* Blood sample for platelets protein analysis (including ACC phosphorylation). After platelets isolation, the remaining plasma will be frozen (2 TUBES CPDA of 8.5 ml).
* Urine sample.

Data collection Data will be collected from Medical Explorer and Q Care, including biological data that are routinely performed in patients admitted in the ICU as platelets count, CRP level, coagulation assessment, renal function and liver enzymology. Follow-up will be performed by at least 3 years and no additional visits will be planned. Events recorded during the follow-up period will be obtained from Medical Explorer and a phone call will be done in case of missing data.

Measurements

* Blood cells count including platelets.
* ACC phosphorylation via western blotting, ECLIA.
* Platelets protein extract for protein acetylation.
* Platelet function ex vivo using Multiplate analysis.
* Plasma sampling.
* Platelets lipidomics analysis. ACC phosphorylation analysis
* Plasma-rich-platelet (PRP) will be obtained after centrifugation. Apyrase and Integrilin are added to limit platelet activation during preparation. PRP will be divided into 3 samples and platelets will be pelleted after centrifugation at 400 g for 10 minutes.
* One of the 3 platelets samples will be lysed with Lemli solution for Western blot analysis of phosphorylated ACC, ACC1 and phosphorylated protein kinase C substrates. All samples will then be stocked at -80°c. In order to compare different immunoblotting, control platelets samples are obtained after thrombin stimulation. Each patient's platelet sample will be compared to the same control sample. The signal of phosphorylated ACC for each patient will be quantified by Image J (Rasband, W.S., ImageJ, U. S. National Institutes of Health, Bethesda, Maryland, USA, http://imagej.nih.gov/ij/, 1997-2014) and will be expressed as a fraction of the control sample signal.
* Level of phosphorylated ACC will be confirmed by electrochemiluminescence (ECLIA, Meso Scale Discovery) and flow cytometry (FACS).
* Protein extracts will be used for platelets protein analysis using immunoblotting.

Plasma sampling

* Coagulation markers including INR, TCA, TT, PTT, Fibrinogen, D-Dimers, Thrombin antithrombin complex (TAT).
* Cytokines measurements (TNF-alpha, IL-1b, IL-6, chemokines- CCL 3, 5, and 18, complement system) as well as inflammatory biomarkers (hypersensitive C-reactive protein).
* Platelets activation biomarkers (sCD62P, sCD40L, CD62P, PF4) (collaboration with Dr C. Oury, GIGA, Université de Liège, Belgium).
* Fibrinolytic biomarkers (u-PA, t-PA and PAI).
* Lipidomic. Urines Samples of urines will be collected in the same times that blood sampling to measure TX2B generation.

Lipidomic analyses Lipidome will be analyzed in collaboration with Christine Des Rosiers in Montréal Heart Insitute. Special attention will be given to metabolites from the COX and LOX pathways (TXA2 and lipoxins).

Sample size

Based on our preliminary data, we determined that enrollment of minimum 46 patients would provide a power of 90% at a significance level of 5% to detect a difference of 0.15 in the phosphorylation of ACC (difference between control group 1 and septic shock population). 20 patients are expected in the exploratory control group.

Covid-19 - Study amendment

Since December 2019, novel Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV- 2) causing Coronavirus disease 2019 (COVID-19) has evolve from an epidemic outbreak in China into a pandemic. Severe infection is mainly responsible for bilateral pneumonia but emerging data indicate that it is a systemic disease involving multiple systems including the hematopoietic and immune system. Endothelial activation, procoagulant state and micro-thrombosis has been shown. However, the pathophysiology has not been demonstrated to be similar to a bacterial sepsis and the above-mentioned metabolic pathway should also be studied in the subgroup of Covid- 19 patients.

Covid-19 group will correspond to patients admitted in the ICU with ARDS due to SARS-Cov-2 infection and PaO2/FiO2 < 200. Inclusion will be done within 5 days after admission and patients with bacterial co-infection will be excluded. We planned to enroll 46 patients, similarly to the control and septic shock group.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent of patients, their relatives or independent physician
* Septic shock defined as a sepsis with vasopressor therapy needed to elevate MAP ≥65 mmHg, and lactate > 2 mmol/L, despite adequate fluid resuscitation of 30mL/kg of intravenous crystalloid within 6 hours. Inclusion within 48 hours of ICU admission.
* Covid-19 patients with ARDS and PaO2/FiO2 < 200. Inclusion within 5 days after ICU admission.

Exclusion Criteria:

* Patients on therapeutic anticoagulation therapy (oral or parenteral) including heparins, fondaparinux, vitamin K antagonist, novel oral anticoagulants, for any reasons DESPITE therapeutic anticoagulation as a treatment for Covid-19 patients.
* Recent (less than 1 month) chemotherapy
* Active inflammatory disease
* Haemophilia and other coagulopathy
* Previous history of thrombocytopenia (<100 000 platelets/mm3)
* Cirrhosis (Child Plug > A)
* Recent (less than 48 hours) major surgery

Exclusion criteria for Covid-19 patients:

- bacterial co-infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Platelets Acetyl-CoA Carboxylase phosphorylation rate | At the time of inclusion
  ACC phosphorylation on Ser79 (phosphoACC) in platelets of patients will be assessed using western blotting. Results will be expressed in arbitrary units (A.U). A signal above 0.5 A.U. has already been shown to be above 2 standard deviation in a healthy population.

SECONDARY OUTCOMES:
Sepsis severity | At the time of inclusion
  Sepsis severity will be assessed using the SOFA score (Sepsis-related Organ Failure Assessment). Range from 0( less severe) to 24 (more severe).
Sepsis severity | At the time of inclusion
  Sepsis severity will be assessed using the APACHE II score) Acute Physiology And Chronic Health Evaluation) Range 0 (less severe) to 299 (more severe).
Mortality rate | 30 days and 1-year follow-up
Platelet function assessment | At the time of inclusion
  Platelet function will be assessed using platelets aggregometry. The Aggregation (in AU), the maximum height of the curve during the measurement period will be assessed.
Platelet function assessment | At the time of inclusion
  Platelet function will be assessed using platelets aggregometry. Area Under the aggregation Curve (AUC) will be assessed and recorded as Units or U.
Platelet function assessment | At the time of inclusion
  Platelet function will be assessed using platelets aggregometry. Velocity (in AU/min), the maximum slope of the curve will be assessed.
Thrombin generation marker rate | At the time of inclusion
  D-Dimers (ng/ml)
Thrombin generation marker rate | At the time of inclusion
  Urinary Thrombin-antithrombin complex (ng/mL)
Tubulin acetylation rate | At the time of inclusion
  Tubulin acetylation will be assessed using western blotting. Results will be expressed in arbitrary units (A.U).
Total platelets lipid content and composition | At the time of inclusion
  Total platelets lipid content and composition will be assessed using metabolomics approach by Mass Spectrometry. Fold-change estimates and corresponding P values were derived from regression models for each lipid species and each predictor. To control for multiple testing, all P values will be further adjusted for Benjamini-Hochberg false discovery rate (FDR), with a FDR <0.05 considered statistically significant
Neutrophils extracellular trap formation | At the time of inclusion
  Myeloperoxidase MPO (ng/mL)
Neutrophils extracellular trap formation | At the time of inclusion
  Citrulinated Histon 3 H3-Cit (ng/mL)
Platelets activation | At the time of inclusion
  Soluble CD62P (ng/mL)
Respiratory failure | At the time of inclusion and through study completion up to day 30
  PaO2/FiO2

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Beauloye, MD, Principal Investigator — Cliniques Universitaires St Luc
Locations (1):
- Cliniques Universitaires St Luc, Brussels, Belgium